CLINICAL TRIAL: NCT07203677
Title: Comparative Effectiveness of Tirzepatide Versus Sitagliptin in Individuals at Cardiovascular Risk (TIRZSITA-CVOT)
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-TIRZSITA
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes Mellitus; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiation of tirzepatide: Exposure group
  Interventions: Drug: Initiation of tirzepatide
- Initiation of sitagliptin: Reference group
  Interventions: Drug: Initiation of sitagliptin

INTERVENTIONS:
Drug: Initiation of tirzepatide — New use of tirzepatide dispensing claim is used as the exposure.
  Groups: Initiation of tirzepatide
Drug: Initiation of sitagliptin — New use of sitagliptin dispensing claim is used as the reference.
  Groups: Initiation of sitagliptin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to assess the comparative effectiveness of tirzepatide vs sitagliptin as a placebo proxy, after the pivotal RCT SURPASS-CVOT (NCT04255433) and its emulation (NCT07088718) demonstrated non-inferiority, leaving both regulators and clinical guideline committees uncertain whether to approve and recommend tirzepatide for a cardiovascular indication. This comparative effectiveness target trial described below draws from eligibility criteria from the SURPASS-CVOT trial and its emulation. Although many features of the target trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the target trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

The purpose of this protocol is to specify the target trial assessing the comparative effectiveness of the dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 receptor agonist (GLP-1-RA) tirzepatide vs the dipeptidyl peptidase-4 inhibitors (DPP4i) sitagliptin on atherosclerotic cardiovascular end points in patients with type 2 diabetes and atherosclerotic cardiovascular disease.

The database study will be a new-user active-comparative study, conducted using 2 national United States claims databases, where we compare the effect of tirzepatide vs sitagliptin in preventing atherosclerotic cardiovascular events. Clinical guidelines during the study period recommended both agents under investigation as second-line options for glucose lowering and were similarly costly.

ELIGIBILITY:
Inclusion Criteria:

* History of MI or stroke, surgical or percutaneous coronary/carotid peripheral artery revascularization, amputation, diagnosis of coronary/carotid/peripheral artery disease
* BMI ≥25.0kg/m2
* Type 2 diabetes
* Age ≥40 years
* Male or female sex

Exclusion Criteria:

* Medullary thyroid carcinoma, MEN syndrome type 2, malignancy
* Treatment for diabetic retinopathy/macular edema, heart failure NYHA IV, gastric emptying abnormality/bariatric surgery, end-stage renal disease or dialysis, pregnancy
* Prior use of pramlintide or any GLP-1-RA except tirzepatide,
* Pancreatitis, liver disease
* Cardiovascular event or intervention, hospitalization for heart failure
* Concurrent use of both drugs i.e. tirzepatide and sitagliptin

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 40 years or older with T2DM and and atherosclerotic cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 49065 (Actual)
Dates: Start 2025-09-19 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin on the composite of myocardial infarction, stroke, or all-cause mortality in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.

SECONDARY OUTCOMES:
Composite of myocardial infarction or stroke | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin on the composite of myocardial infarction or stroke in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
Myocardial infarction | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin at preventing myocardial infarction in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
Stroke | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin at preventing stroke in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
All-cause mortality | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin at preventing all-cause mortality in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
Composite of myocardial infarction, stroke, coronary revascularization, or hospitalization for unstable angina. | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin on the composite of myocardial infarction, stroke, coronary revascularization, or hospitalization for unstable angina in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
Serious bacterial infections | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin on the safety outcome of serious bacterial infections in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
Urinary tract infections | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin on the safety outcome of urinary tract infections in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.
Gastrointestinal adverse events | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs sitagliptin on the safety outcome of gastrointestinal adverse events in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.

OTHER OUTCOMES:
Hernia and lumbar radiculopathy | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs sitagliptin on negative control outcomes, including (1) hernia and (2) lumbar radiculopathy in patients with type 2 diabetes and atherosclerotic cardiovascular disease when following the inclusion and exclusion criteria of the SURPASS-CVOT trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Amendment 2 to Study Protocol with Statistical Analysis Plan (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT07203677/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Amendment to Study Protocol with Statistical Analysis Plan (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT07203677/Prot_SAP_001.pdf
  • Study Protocol: Study Protocol with Statistical Analysis Plan (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT07203677/Prot_000.pdf